CLINICAL TRIAL: NCT00249548
Title: Low-Cost Contingency Management for Hispanic Outpatients
Brief Title: Low-Cost Contingency Management for Hispanic Outpatients - 3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: UConn Health (Other)
Responsible Party: Nancy Petry, Ph.D., UConn Health Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NIDA-13444-3; R01-13444-3
Record Dates: First submitted 2005-11-03; First posted 2005-11-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-05

CONDITIONS: Substance Abuse
Keywords: contingency management; substance abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Contingency management

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a lower-cost contingency management (CM) procedure in Hispanic substance abusing outpatients. Thirty individuals meeting DSM-IV criteria for substance dependence receive one of two conditions: (a) standard treatment, or (b) standard treatment plus prize CM. Using a cross-over design, CM is implemented in a community-based outpatient clinic and compared with non-CM in the same clinic. The participating clinic is randomly assigned to receive either the CM or non-CM phase first; 15 weeks after the final participant in one phase is enrolled, a one-week washout period occurs, followed by a switch to the other phase. Patients initiating outpatient treatment during the non-CM phase receive standard treatment and submit urine and breath samples 2/week during Weeks 1-6 and 1/week during Weeks 7-12. Patients initiating treatment during the CM phase also receive standard treatment and the same breath and urine monitoring. In addition, they earn the opportunity to win prizes for coming to treatment and for submitting negative breath and urine samples. Follow-up interviews are conducted at 1,3,6 and 9 months following intake during which substance use and psychosocial functioning are assessed.

ELIGIBILITY:
Inclusion criteria:

* age > 18 years
* current DSM-IV substance dependence.

Exclusion criteria:

* have a serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, bipolar disorder, severe or psychotic major depression, or suicide risk) on the basis of history or medical examination
* have dementia (<23 on the Mini Mental State Exam; Folstein et al. 1975)
* DSM-IV diagnosis of pathological gambling
* plans to move from the Hartford are within 9 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-08; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Drug use | baseline and each follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Petry, Ph.D., Principal Investigator — UConn Health